CLINICAL TRIAL: NCT06375057
Title: Relationship Between Acute Phase Markers and Acute Post-operative Pain in Laparoscopic Cholecystectomy: An Observational Study
Brief Title: Relationship Between Acute Phase Markers and Post-operative Pain in Laparoscopic Cholecystectomy: An Observational Study
Status: Recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Augusto Lauro, Associate professor, University of Roma La Sapienza
Other Study IDs: asiamkfv49wurfpylld2m6g7cr4kz6
Record Dates: First submitted 2024-04-11; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing laparoscopic cholecystectomy
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — A blood sample is taken the day after surgery

SUMMARY:
Many patients undergoing laparoscopic cholecystectomy are prone to developing acute and chronic post-operative pain.

The aim of the study is to show a possible correlation between pain and acute phase proteins in order to:

* predict the severity of pain;
* select most suitable pain relief therapy for the patient.

DETAILED DESCRIPTION:
The day after surgery, some serum markers are determined by a blood sample.

The markers analyzed are:

* Leukocytes;
* C-reactive protein (CRP);
* D-dimer;
* Fibrinogen;
* Neutrophil-to-Lymphocyte Ratio (NLR).

Pain level is assessed using the NRS scale at different times:

* 1st post-operative day;
* 7th post-operative day;
* One month after surgery;
* Three months after surgery;
* Six months after surgery.

Other data collected for the study are: gender, age, BMI.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes patients undergoing laparoscopic cholecystectomy
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relationship Between Post-operative Pain and C Reactive Protein (CRP) in Laparoscopic Cholecystectomy | one day
  The study compares post-operative pain, measured with the NRS scale, with CRP (µg/L) levels 24 hours after surgery
Relationship Between Post-operative Pain and D-dimer in Laparoscopic Cholecystectomy | one day
  The study compares post-operative pain, measured with the NRS scale, with D-dimer (µg/L FEU) levels 24 hours after surgery
Relationship Between Post-operative Pain and Fibrinogen in Laparoscopic Cholecystectomy | one day
  The study compares post-operative pain, measured with the NRS scale, with fibrinogen (g/L) levels 24 hours after surgery
Relationship Between Post-operative Pain and white blood cell count in Laparoscopic Cholecystectomy | one day
  The study compares post-operative pain, measured with the NRS scale, with white blood cell count (x 10^9/L) 24 hours after surgery
Relationship Between Post-operative Pain and Neutrophil to Lymphocyte Ratio (NLR) in Laparoscopic Cholecystectomy | one day
  The study compares post-operative pain, measured with the NRS scale, with Neutrophil to Lymphocyte Ratio (NLR) 24 hours after surgery. NLR results from the ratio between the level of neutrophils and lymphocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusto Lauro, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rathee A, Chaurasia MK, Singh MK, Singh V, Kaushal D. Relationship Between Pre- and Post-Operative C-Reactive Protein (CRP), Neutrophil-to-Lymphocyte Ratio (NLR), and Platelet-to-Lymphocyte Ratio (PLR) With Post-Operative Pain After Total Hip and Knee Arthroplasty: An Observational Study. Cureus. 2023 Aug 20;15(8):e43782. doi: 10.7759/cureus.43782. eCollection 2023 Aug. PMID 37731439
- [Background] Shu B, Xu F, Zheng X, Zhang Y, Liu Q, Li S, Chen J, Chen Y, Huang H, Duan G. Change in perioperative neutrophil-lymphocyte ratio as a potential predictive biomarker for chronic postsurgical pain and quality of life: an ambispective observational cohort study. Front Immunol. 2023 Apr 12;14:1177285. doi: 10.3389/fimmu.2023.1177285. eCollection 2023. PMID 37122722
- [Background] Gonzalez-Callejas C, Aparicio VA, De Teresa C, Nestares T. Association of Body Mass Index and Serum Markers of Tissue Damage with Postoperative Pain. The Role of Lactate Dehydrogenase for Postoperative Pain Prediction. Pain Med. 2020 Aug 1;21(8):1636-1643. doi: 10.1093/pm/pnz325. PMID 31845982

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT06375057/Prot_SAP_000.pdf